CLINICAL TRIAL: NCT03584035
Title: Effects of Sensorimotor Integration Exercises on Balance and Fall Efficacy in Sub-acute Stroke
Brief Title: Sensorimotor Integration Exercises on Post-stroke Balance and Fall Efficacy
Acronym: SMIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of Medical Technology, Yangon (Other)
Responsible Party: Principal Investigator, Thin Thin Moe, Ph D, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2018
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: sensory motor integration exercise
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will do all assessments (pre and post intervention) without group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory motor integration group (Experimental): Sensory-motor integration exercises with 3 progressive steps, 30 minutes per sessions, 3 sessions per week for 6 weeks.
  Interventions: Behavioral: sensory motor integration exercises
- Conventional group (Active Comparator): Conventional exercises include simple passive and active exercises and lower extremities strengthening exercises for balance and ambulation. The exercise session will last 30 minutes for 3 sessions per week. The total intervention period is 6 weeks.
  Interventions: Behavioral: conventional physiotherapy

INTERVENTIONS:
Behavioral: sensory motor integration exercises — Sensorimotor integration exercises will be given in study group. The exercises will be performed in standing, sitting and walking. Exercises will be progressively increased from eye open to closed , floor to mat and head turns to right & left under the supervision of physiotherapist. Sensorimotor integration exercises will take 45 minutes in each session.
  Arms: Sensory motor integration group
Behavioral: conventional physiotherapy — Conventional physiotherapy will take 30 minutes in each session, taking three sessions per weeks for six weeks. The exercises include simple lower extremity exercise and ambulatory training such as sit to stand, stepping, lateral and backward walking, and tandom walking etc.
  Arms: Conventional group

SUMMARY:
To study the effect of sensorimotor integration exercises on balance and fall efficacy in sub-acute stroke by performing 18 balance training exercises with three progressive steps.

DETAILED DESCRIPTION:
Balance impairment after stroke is significantly correlated with fall risk. To improve balance and reduce fall efficacy, the participants in the study group will be trained by six weeks three progressive steps of sensorimotor integration exercises. Each exercise step will take 30 minutes of a practice session, three sessions per week. Conventional physiotherapy (passive and active exercises and lower extremities strengthening exercises) will be given to the control group. The changes in balance performance and fall efficacy will be measured and compared within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* First episode of sub-acute stroke (from 1 to 26 weeks) referred from physicians
* Both sexes
* Age above 20
* Good cognition (Mini Mental State Examination Scale ≥24)
* Moderate and moderately severe disability (Modified Rankin Scale- 3 and 4)
* Impaired balance (BBS <41)

Exclusion Criteria:

* Recurrent stroke
* Associated with other neurological conditions (such as Parkinson's disease, Epilepsy, meningitis)
* Deficits of somatic sensation involving the paretic limb (Fugl-Meyer Assessment - sesation< 1)
* Lower extremity weight bearing pain (Fugl-Meyer Assessment- pain <1)
* Low back pain (VAS ≥ 3)
* Severe visual deficits which cannot be corrected by lens or glasses
* Symptomatic vestibular disorders (Paroxysmal postural vertigo)
* Associated serious cardiac disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 6 weeks
  14 items to measure static and dynamic balance

SECONDARY OUTCOMES:
Functional Reach Test | 6 weeks
  To assess the stability by measuring the maximum distance while standing in a fixed position
Fall Efficacy Scale | 6 weeks
  Short, easy questionnaire that provides information about how much fear of fall, which is comprised of 16-items concerning confidence in maintaing balance during activities.

CONTACTS AND LOCATIONS:
Overall Officials: May Phyu Phyu Maung, B.Med.Tech, Principal Investigator — University of Medical Technology, Yangon; Thin Thin Moe, Ph.D, Principal Investigator — Mahidol University; Myo Thuzar Khin, Ph.D, Study Chair — University of Medical Technology, Yangon
Locations (2):
- Burma (2):
  - National Rehabilitation Hospital, Yangon
  - Physical Medicine and Rehabilitation Department, Yangon General Hospital, Yangon